CLINICAL TRIAL: NCT07063329
Title: An Open-label, Multicenter Phase Ib/II Clinical Study to Evaluate the Safety, Efficacy, and Pharmacokinetic of PLB1004 Capsules Combined With Platinum-based Doublet Chemotherapy in Patients With EGFR Mutation-positive NSCLC
Brief Title: Phase I/II Study of PLB1004 Combined With Platinum-based Doublet Chemotherapy in Patients With EGFR Mutation-positive
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avistone Pharmaceutical（Ningbo）Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLB1004 +Chemo-NSCLC-Ib/II-01
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- phase Ib Dose Escalation (Experimental)
  Interventions: Drug: PLB1004 80mg/160mg/240mg oral once daily Combined with Platinum-Based Chemotherapy
- phase Ib Dose Expansion (Experimental)
  Interventions: Drug: PLB1004 80mg/160mg/240mg oral once daily Combined with Platinum-Based Chemotherapy
- phase II Cohort1 (Experimental)
  Interventions: Drug: RP2D of PLB1004 oral once daily Combined with Platinum-Based Chemotherapy
- phase II Cohort2 (Experimental)
  Interventions: Drug: RP2D of PLB1004 oral once daily Combined with Platinum-Based Chemotherapy

INTERVENTIONS:
Drug: PLB1004 80mg/160mg/240mg oral once daily Combined with Platinum-Based Chemotherapy — For non-squamous NSCLC patients：Pemetrexed (500 mg/m2) plus carboplatin (AUC5) or cisplatin（75 mg/m²）on Day 1 of 21day cycles (every 3 weeks) , followed by PLB1004 80mg/160mg/240mg oral once daily。 For squamous NSCLC subjects: Docetaxel（75 mg/m² ）or paclitaxel（175 mg/mg） plus carboplatin (AUC5) or cisplatin（75 mg/m²）on Day 1 of 21day cycles (every 3 weeks) , followed by PLB1004 80mg/160mg/240mg oral once daily.
  Arms: phase Ib Dose Escalation
Drug: PLB1004 80mg/160mg/240mg oral once daily Combined with Platinum-Based Chemotherapy — Multiple doses of PLB1004 for oral administration. Platinum-based chemotherapy is combined and administered on Day 1 of 21days（every 3 weeks).
  Arms: phase Ib Dose Expansion
Drug: RP2D of PLB1004 oral once daily Combined with Platinum-Based Chemotherapy — RP2D of PLB1004 as determined during Phase Ib . Platinum-based chemotherapy is combined and administered on Day 1 of 21days（every 3 weeks）.
  Arms: phase II Cohort1
Drug: RP2D of PLB1004 oral once daily Combined with Platinum-Based Chemotherapy — RP2D of PLB1004 as determined during Phase Ib，patients will undergo surgical treatment after 3 cycles of combination therapy with platinum-based chemotherapy. Post-surgery, they will receive an additional cycle of platinum-based chemotherapy followed by 13 cycles of maintenance therapy with PLB1004.
  Arms: phase II Cohort2

SUMMARY:
Tyrosine Kinase Inhibitor (TKI) that targets Epidermal Growth Factor Receptor (EGFR) mutations. Unfortunately, despite the benefit observed for patients treated with EGFR-TKI, the vast majority of cancers are expected to develop resistance to the drug over time. The exact reasons why resistance develops are not fully understood but based upon clinical research it is hoped that combining PLB1004 with another type of anti-cancer therapy known as chemotherapy will delay the onset of resistance and the worsening of a patient's cancer.

In recent years, clinical studies on the combination of EGFR-TKI and chemotherapy have made important progress, suggesting that the combination of EGFR-TKI and chemotherapy further enhances the therapeutic benefit in EGFR-mutant positive NSCLC.

Both preclinical and clinical data indicate that PLB1004 exhibit good antitumor activity and relatively durable efficacy in NSCLC patients with EGFR mutations. They can reduce tumor burden, control tumor progression, and improve the survival benefit of patients, which is expected to provide an effective treatment option for such patients.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, dose-escalation and dose-expansion Ib/II phase study, aiming to evaluate the clinical safety, tolerability, PK and preliminary efficacy of PLB1004 combined with platinum-based doublet chemotherapy in NSCLC patients with EGFR mutations. The study consists of two parts: the phase Ib dose-escalation study and dose-expansion study, as well as the phase II clinical study. The target population of the phase Ib study is patients with confirmed locally advanced or metastatic NSCLC harboring EGFR mutations who have received or not received systemic antitumor therapy. The II phase clinical study sets up two cohorts. Cohort 1: patients with confirmed locally advanced or metastatic NSCLC harboring EGFR mutations who have received or not received systemic antitumor therapy; Cohort 2: patients with newly diagnosed resectable stage II-III NSCLC harboring EGFR mutations who have not received systemic antitumor therapy. A total of 79-108 patients are planned to be enrolled in the study, which is divided into a screening period, a treatment period and a follow-up period. During the administration of the study drug, follow-up will be conducted every 6 weeks in the first year and every 12 weeks from the second year onwards.

ELIGIBILITY:
Inclusion Criteria:

* 1. Phase Ib Dose-escalation Part : Patients with histologically or cytologically confirmed unresectable locally advanced (stage IIIB and IIIC) or metastatic (stage IV) NSCLC (according to the eighth edition of the AJCC lung cancer staging criteria) who have disease progression or intolerance after previous systemic treatment. Specific treatment requirements are as follows:

  * Patients with EGFR sensitive mutations: They must have received EGFR-TKI treatment. If only first/second-generation EGFR-TKIs were used, T790M negativity must be confirmed.
  * Patients with other EGFR mutations such as EGFR exon 20 insertion: They must have received platinum-based chemotherapy.

Phase Ib Dose-expansion part and Cohort 1 of Phase II: Patients with histologically or cytologically confirmed unresectable locally advanced (stage IIIB and IIIC) or metastatic (stage IV) NSCLC (according to the eighth edition of AJCC staging) who have not received previous systemic treatment or have received systemic treatment.

Cohort 2 of Phase II: Patients with histologically confirmed resectable stage II-III NSCLC (according to the eighth edition of AJCC staging) who have not received previous systemic treatment; among them, N2 is defined as single-station mediastinal lymph node non-bulky metastasis (lymph node short diameter <2 cm) confirmed by imaging and pathology, with expected complete resection.

* 2. Previous tumor tissue or pleural effusion or blood sample confirmed positive for EGFR mutation.
* 3. Measurable lesions at baseline according to RECIST 1.1 criteria.
* 4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
* 5. Estimated life expectancy is more than 12 weeks.
* 6. It has been medically evaluated and determined that the organ functions are good (within 7 days before the first study drug administration), including:

  * hematological : absolute neutrophil count (ANC) ≥ 1.5 × 109/L, hemoglobin ≥ 90 g/L, platelets ≥ 100 × 109/L. Platelet transfusion is not allowed within 3 days before testing, red blood cell transfusion is not allowed within 14 days before testing, and hematopoietic growth factor therapy is not allowed within 7 days before testing (pegylated granulocyte colony-stimulating factor [G-CSF] or erythropoietin [EPO] is within 14 days before testing).
  * liver function: serum TBIL ≤ 1.5×ULN (in patients with known Gilbert syndrome, TBIL ≤ 3×ULN and direct bilirubin [DBIL] ≤ 1.5×ULN), serum ALT/AST ≤ 2.5×ULN (for patients with confirmed liver metastases, ≤ 5.0×ULN).
  * Renal function: Creatinine clearance ≥ 50 mL/min.
  * coagulation function, defined as (including during anticoagulant therapy): prothrombin time (PT)<1.5 × ULN, activated partial thromboplastin time (APTT)<1.5 × ULN. If the subject is receiving anticoagulant therapy, they must receive a stable dose of anticoagulant at least one month prior to the first study administration.
* 7. For cohort 2 of phase II: According to the surgeon's assessment, the total lung function can tolerate the planned pulmonary resection surgery.
* 8. Female patients must use effective contraceptive measures during the study and for 90 days after the end of study treatment, and must not breastfeed.Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to the first dose.

Exclusion Criteria:

* 1. Participated in other therapeutic clinical trials within 28 days prior to the first dose。
* 2. Patients underwent major organ surgery within 4 weeks prior to the first dose.or is expected to undergo major surgery during the study.
* 3. Have received lung field or whole-brain radiotherapy within 28 days before the first study drug administration, or has received palliative local radiotherapy within 14 days before the first dose。
* 4. Patients received antitumour traditional Chinese medicine within 1 weeks prior to the first dose，and received local anti-tumor drug therapy (such as thoracic or abdominal perfusion, etc.) within 14 days or within 5 half-lives (whichever is shorter)。
* 5. Patients with malignancies other than tumors treated in this study (except: malignancies that are cured and have not recurred within 3 years prior to study entry; completely resected basal cell and squamous cell skin cancer; completely resected carcinoma in situ of any type).
* 6. Adverse effects of previous anti-tumor therapy have not recovered to CTCAE 5.0 grade rating of ≤ grade 1 (except for toxicity judged by the investigator be of no safety risk, such as alopecia, skin pigmentation, etc.)
* 7. Have received systemic administration of potent inhibitors/inducers of CYP3A4 within 7 days prior to the first dose of treatment/randomization or are expected to receive systemic administration of these drugs during study treatment.
* 8. Patients have symptomatic central nervous system (CNS) metastases, meningeal metastases, or a primary CNS tumor that is associated with progressive neurological symptoms.
* 9. Patients have a history of severe cardiovascular disease, including but not limited to:

  * Mean QT interval corrected using Fridericia's formula (QTcF) from three times> 480ms at rest.
  * New York Heart Association (NYHA) ≥ class II heart failure or left ventricular ejection fraction (LVEF) < 50%.
* 10. Hypertension remains uncontrolled（systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg ） after aggressive antihypertensive therapy.
* 11. Patients with active uncontrolled systemic bacterial, viral, or fungal infection despite optimal treatment Active hepatitis (Hepatitis B: HBsAg-positive and HBV-DNA ≥ 2000 IU/ mL; Hepatitis B: HCV antibody-positive , HIV antibody-positive; Active syphilis, the onset period of keratitis or ulcerative keratitis.
* 12. Patients are unable to swallow the drug orally, or has a condition that seriously affects gastrointestinal absorption in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2028-03-08 (Estimated); Study Completion 2028-07-08 (Estimated)

PRIMARY OUTCOMES:
Phase Ib： Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 12 months
  To evaluate the tolerability and safety of PLB1004 combined with platinum-based doublet chemotherapy in patients with epidermal growth factor receptor (EGFR) mutation positive NSCLC
Phase Ib： Incidence of dose-limiting toxicities (DLT) as defined in the protocol | 12 months
  To determine the maximum tolerated dose (MTD) and/or dose-limiting toxicities (DLT) of combination therapy of PLB1004 combined with platinum-based doublet chemotherapy in patients with EGFR mutation positive NSCLC
Phase Ib： Recommended Phase II Dose (RP2D) | 12 months
  To determine the recommended phase II dose (RP2D) of PLB1004 in combination with platinum-based doublet chemotherapy in subjects with EGFR mutation positive NSCLC
Phase Ib： Overall Response Rate (ORR） | 24 months
  ORR is defined as the proportion of subjects with confirmed best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1
Phase II： To evaluate the efficacy of PLB1004 in combination with platinum-based doublet chemotherapy at the RP2D in subjects with EGFR mutation positive locally advanced or metastatic NSCLC | 36 months
  Objective response rate (ORR) as evaluated by the investigator according to RECIST v1.1
Phase II： To evaluate the efficacy of PLB1004 in combination with platinum-based doublet chemotherapy at the RP2D RP2D in newly diagnosed resectable stage II-III NSCLC subjects with EGFR mutation positive | 12 months
  Major pathological response (MPR) evaluated by the blinded independent pathology review committee (BIPR)

SECONDARY OUTCOMES:
Cmax | 12 months
  Single-dose PK parameters: Peak concentration (Cmax)
DOR | 36 months
  Duration of response (DoR)
PFS | 36 months
  Progression-Free Survival
Tmax | 12 months
  Time to peak concentration (Tmax)
(AUC0-t） | 12 months
  Evaluation of the area under the concentration-time curve (AUC0-t)
T 1/2 | 12 months
  Assessment of the first dose elimination half-life (T 1/2)
CL/F | 12 months
  Assessment of apparent clearance rate of the first dose (CL/F)
Vz/F | 12 months
  Apparent volume of distribution
DCR | 36 months
  Disease Control Rate
OS | 36 months
  Overall Survival
EFS | 36 months
  Event-Free Survival
pCR | 36 months
  pathological Complete Response
DFS | 36 months
  Disease-Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu M.D, Ph.D., Principal Investigator — Shanghai Chest Hospital; Deng Hou Master, Study Director — Avistone Pharmaceutical（Ningbo）Co., LTD.
Locations (1):
- Shanghai Chest hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No